CLINICAL TRIAL: NCT06331104
Title: Treatment of Giant Cell Bone Tumor With Purerin: New Insights From Network Pharmacology, Bioinformatics Analysis, and Experimental Verification
Brief Title: Network Pharmacology Prediction: Mechanism Study of Puerarin in the Treatment of Giant Cell Tumors of Bone
Status: Completed | Type: Observational
Sponsor: Changye Zou (Other)
Responsible Party: Sponsor-Investigator, Changye Zou, Department of Orthopedic Oncology, The First Affiliated Hospital of Sun Yat-sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: ChangyeZou
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Giant Cell Tumors
Keywords: Giant Cell Tumors; Puerarin; Treatment; Traditional Chinese medicine; Network Pharmacology
MeSH Terms: conditions — Giant Cell Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Immunohistochemistry (IHC) and immunofluorescence staining were performed on the GCTB tissues of 145 patients (2 normal tissues, 51 recurrent, and 92 primary) from the First Affiliated Hospital of Sun Yat sen University to verify the differential expression and distribution of P27 and ESR1 in recurrent and primary lesions of giant cell tumor of bone patients. One patient's tissue was used for transcriptome sequencing to analyze changes in gene expression levels before and after routine treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P27 expression groups: 12 immunohistochemical sections were scored under the microscope (staining intensity scores: negative 0 points, weak 1 point, medium 2 points, strong 3 points; positive cell frequency scores: less than 5% 0 points, 2-25% 1 point, 26-50% 2 points, 51-75% 3 points, greater than 75% 4 points).
  Interventions: Genetic: gene expression levels
- ESR1 expression groups: 12 immunohistochemical sections were scored under the microscope (staining intensity scores: negative 0 points, weak 1 point, medium 2 points, strong 3 points; positive cell frequency scores: less than 5% 0 points, 2-25% 1 point, 26-50% 2 points, 51-75% 3 points, greater than 75% 4 points).
  Interventions: Genetic: gene expression levels

INTERVENTIONS:
Genetic: gene expression levels — 12 immunohistochemical sections were scored under the microscope (staining intensity scores: negative 0 points, weak 1 point, medium 2 points, strong 3 points; positive cell frequency scores: less than 5% 0 points, 2-25% 1 point, 26-50% 2 points, 51-75% 3 points, greater than 75% 4 points).

SUMMARY:
Based on network pharmacology analysis, this study aims to explore the potential therapeutic targets and molecular mechanisms of puerarin on giant cell tumor of bone (GCTB) genes.

DETAILED DESCRIPTION:
The giant cell tumor of bone's pathological genes were discovered from DisGeNET and GeneCards databases. The therapeutic genes of puerarin were gathered from Swiss Target Prediction, CTD(Comparative Toxicogenomics Database), PharmMapper, and TCMSP databases (Traditional Chinese Medicine Systems Pharmacology Database and Analysis Platform). Cytoscape software was used with the MCODE algorithm to calculate key potential therapeutic targets of puerarin against GCTB. The bulk RNA-seq datasets (GSE102193) were used to identify differential expression of potential therapeutic genes. The sc RNA-seq (GSE168664) was utilized to determine the expression distribution of different cell clusters. Essential targets of puerarin against GCTB underwent function and pathway enrichment assays to elucidate biological processes and signaling pathways. Furthermore, the investigators conducted a comparison to determine if the primary biological processes and pathways following denosumab treatment exhibit resemblances to the potential mechanisms of puerarin action. Molecular docking and dynamics simulation were conducted to evaluate interactions between selected potential therapeutic targets and puerarin. Immunohistochemical (IHC) and immunofluorescence (IF) staining were performed to identify the expression of crucial markers in human GCTB tissue. Expression levels of pivotal genes in primary BMSC cells and primary GCTB cells and their alteration following puerarin treatment in primary GCTB cells were evaluated.The significance of differences between groups was estimated by the Student t-test or Wilcoxon test. In all the statistical analyses, data with two-tailed p < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as a patient with giant cell tumor of bone;
2. Performing surgical treatment in 1st hospital of SYSU;
3. Having complete clinical registration information;
4. Preserve surgical or puncture specimens;

Exclusion Criteria:

1. Non bone giant cell tumor patients;
2. No surgical treatment was performed;
3. Incomplete clinical information registration;
4. No preserved surgical or puncture specimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1st hospital of SYSU provides diagnosis and treatment that meets the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2012-06-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
P27 expression levels | 2023-05-18 - 2023-08-31
  12 immunohistochemical sections were scored under the microscope (staining intensity scores: negative 0 points, weak 1 point, medium 2 points, strong 3 points; positive cell frequency scores: less than 5% 0 points, 2-25% 1 point, 26-50% 2 points, 51-75% 3 points, greater than 75% 4 points).
ESR1 expression levels | 2023-05-18 - 2023-08-31
  12 immunohistochemical sections were scored under the microscope (staining intensity scores: negative 0 points, weak 1 point, medium 2 points, strong 3 points; positive cell frequency scores: less than 5% 0 points, 2-25% 1 point, 26-50% 2 points, 51-75% 3 points, greater than 75% 4 points).

CONTACTS AND LOCATIONS:
Overall Officials: Changye Zou, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Churong Yan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets are available from the corresponding author (zouchy@mail.sysu.edu.cn) on reasonable request after SCI online.
Supporting Information: Study Protocol, SAP
Time Frame: SCI online. The datasets are available from the corresponding author on reasonable request.
Access Criteria: The datasets are available from the corresponding author (zouchy@mail.sysu.edu.cn) on reasonable request after SCI online.